CLINICAL TRIAL: NCT04436588
Title: DDX3X Related Disorder : Clinical Phenotype, Neuropsychological Profile and Epigenetic Signature.
Brief Title: Better Delineation of DDX3X Related Phenotype and Epigenetic Signature.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Association Xtraordinaire sub-group DDX3X (Unknown); Genida (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0353
Record Dates: First submitted 2020-06-10; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Intellectual Developmental Disorder; X-LINKED
Keywords: DDX3X; Syndromic; SNIJDERS BLOK
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DDX3X: DDX3X
  Interventions: Genetic: Epigenetic signatures

INTERVENTIONS:
Genetic: Epigenetic signatures — Epigenetic signatures (Dr Sadikovic' lab, London, Ontario, Canada)

SUMMARY:
DDX3X related disorder is mainly characterised by developmental delay (DD) and intellectual disability (ID), ranging from mild to severe, and neuroimaging abnormalities.

The aims of this study are first to better delineate the clinical phenotype, as well as the neuropsychological profile and, second, to study the epigenetic signature in a cohort of individuals with DDX3X pathogenic variants. This work will conduct to a MD thesis of a clinical resident geneticist in France.

Physician that will participate will fill an Excel sheet regarding the clinical and neuropsychological assessment. The investigators will be also happy to have a DNA sample with a minimum 0.5ug of peripheral blood genomic DNA. The investigators will gather the DNA in Montpellier genetic lab (Dr Mouna BARAT) and send the batch to the Dr Sadikovic' lab.

Between 2018 and 2020, the investigators have already recruited data from individuals with DDX3X pathogenic variants from several European and Asian genetic centres

DETAILED DESCRIPTION:
The investigators aim to better understand and delineate the genetic syndrome DDX3X.

This genetic disorder was described in 2015 by Lot Snijders Blok et al. (DOI https://doi.org/10.1016/j.ajhg.2015.07.004:).

Since this first publication of 38 female individuals carrying a pathogenic mutation DDX3X, 15 more individuals have been reported.

The investigators are seeking to better define the phenotype of individuals with pathogenic variants of DDX3X, to better understand intellectual functioning as well as the strengths and weaknesses of intellectual functioning by collecting standardized neuropsychological assessments already performed such as WPPSI/WISC and WAIS. For this purpose, the investigators will gather clinical and neuropsychological data already carried out in the context of care.

Finally, the investigators will attempt to identify an epigenetic signature in this genetic disease. To this end, the investigators will collect genomic DNA from peripheral blood already collected for genetic analysis and send an anonymized batch of samples to our collaborator, Dr. Bekim Sadicovik. Dr. Bekim Sadicovik and his team will compare the epigenetic DNA methylation-type markers with the corresponding sex and age controls. If specific probes are abnormally methylated in DDX3X individuals, this will determine a disease-specific epigenetic signature. The investigators will then be able to propose an epigenetic signature for individuals with uncharacterized DDX3X variations (class 3, VUS). This method will make it possible to define whether the variation is responsible for the disease or not without going through functional analysis steps that are difficult to implement routinely.

The expected benefits are a better understanding of DDX3X disease, keys to neuropsychological rehabilitation, a better understanding of human brain functions, the possibility of proposing an epigenetic signature for people in whom it is not possible to decide whether a variation in the DDX3X gene is pathological or not

ELIGIBILITY:
Inclusion criteria:

- DDX3X pathogenic Variant

Exclusion criteria:

* no pathogenic variant in DDX3X
* no consent for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with DDX3X pathogenic Variant
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological phenotype will be assessed using Wechsler scales | 1 day
  DDX3X related clinical and neuropsychological phenotype. Neuropsychological phenotype will be assessed using Wechsler scales. The phenotype of individuals will be assessed using a questionnaire sent to their geneticist
Measurement and comparison of the methylation of the cpg sites" | 1 day
  Epigenetic signature will be investigated by measurement and comparison of the methylation of the cpg sites

CONTACTS AND LOCATIONS:
Overall Officials: David GENEVIEVE, Principal Investigator — Department of Medical Genetics
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC